CLINICAL TRIAL: NCT07059975
Title: UPdated Disease Monitoring And Treatment for Enhanced Outcomes for Pediatric AML: A Pilot Trial
Brief Title: UPDATE AML: UPdated Disease Monitoring And Treatment for Enhanced Outcomes for Pediatric AML
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Joanna Yi (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor-Investigator, Joanna Yi, Associate Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-56184 UPDATE AML
Record Dates: First submitted 2025-06-18; First posted 2025-07-11 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia; Pediatric AML
Keywords: venetoclax; measurable residual disease (MRD); digital PCR
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm, Residual | interventions — Idarubicin; fludarabine; Cytarabine; venetoclax; Etoposide; asparaginase erwinia chrysanthemi recombinant

STUDY DESIGN:
Intervention Model Description: Pilot study with assigned risk-based treatment arms, all receiving the study interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Intermediate Risk (IR) AML (Experimental): Patients will receive Ida-FLA as Induction 2, cytarabine/etoposide ("AE") as Intensification 1, VIA as Intensification 2, and Capizzi AraC as intensification 3.
  Interventions: Drug: Idarubicin Hydrochloride; Drug: Fludarabine; Drug: Cytarabine (Ara-C); Drug: Venetoclax; Drug: Etoposide; Drug: Asparaginase Erwinia Chrysanthemi (recombinant); Drug: Intrathecal triple
- High risk (HR) AML (Experimental): Patients will receive Ida-FLA as Induction 2 and VIA as Intensification 1. These patients will then proceed on to a hematopoietic stem cell transplantation if an appropriate donor is found, otherwise will receive 2 more cycles of chemotherapy following the IR regimen.
  Interventions: Drug: Idarubicin Hydrochloride; Drug: Fludarabine; Drug: Cytarabine (Ara-C); Drug: Venetoclax; Drug: Intrathecal triple
- Low risk (LR) (Other): Low risk pediatric AML patients will receive standard of care chemotherapy but have the option to participate in correlative studies
  Interventions: Other: SOC

INTERVENTIONS:
Drug: Idarubicin Hydrochloride — Idarubicin is given in combination with fludarabine and cytarabine for Ida-FLA, and in combination with venetoclax and cytarabine for VIA.
  Arms: High risk (HR) AML; Intermediate Risk (IR) AML
Drug: Fludarabine — Fludarabine is given in combination with idarubicin and cytarabine for Ida-FLA.
  Arms: High risk (HR) AML; Intermediate Risk (IR) AML
Drug: Cytarabine (Ara-C) — Cytarabine is given in combination with other chemotherapy agents in every cycle and both arms.
  Arms: High risk (HR) AML; Intermediate Risk (IR) AML
Drug: Venetoclax — Venetoclax is given in combination with idarubicin and cytarabine for VIA.
  Arms: High risk (HR) AML; Intermediate Risk (IR) AML
Drug: Etoposide — Etoposide is given in combination with cytarabine for AE, as Intensification 1 for IR patients.
  Arms: Intermediate Risk (IR) AML
Drug: Asparaginase Erwinia Chrysanthemi (recombinant) — Rylaze is given in combination with cytarabine for Intensification 3 for IR patients.
  Arms: Intermediate Risk (IR) AML
Drug: Intrathecal triple — Methotrexate, hydrocortisone and cytarabine are combined into one preparation for intrathecal administration at multiple time points during treatment.
  Arms: High risk (HR) AML; Intermediate Risk (IR) AML
Other: SOC — Low-Risk Patients will receive Texas childern's Hospital practice standard for de novo AML.
  Arms: Low risk (LR)

SUMMARY:
This research study investigates the tolerability of substituting two cycles of chemotherapy into the standard pediatric acute myeloid leukemia (AML) chemotherapy treatment regimen for patients with newly diagnosed AML at intermediate-risk (IR) and high-risk (HR) of relapse. The goal is to achieve similar or better survival with chemotherapy cycles that are intensive but less likely to cause long-term complications. Patients will enroll on this trial at the end of their first induction cycle.

The two cycles to be substituted are:

* "Ida-FLA" (idarubicin+fludarabine/cytarabine) as Induction 2
* "VIA" (venetoclax+idarubicin+cytarabine) as Intensification 1 of the HR treatment regimen, and Intensification 2 of the IR treatment backbone.

Researchers will evaluate side effects and outcomes for up to three years after enrollment.

Participants will also have the opportunity to participate in optional research studies including patient surveys and blood and bone marrow sample testing.

DETAILED DESCRIPTION:
UPDATE AML is a research study that investigates the tolerability of substituting two cycles of chemotherapy into the standard pediatric acute myeloid leukemia (AML) chemotherapy treatment regimen for patients at intermediate-risk (IR) and high-risk (HR) of the leukemia coming back ("relapse"). Newly diagnosed patients will receive standard Induction 1 treatment off study. If they do not have a FLT3-ITD mutation, they will be eligible to complete treatment on the UPDATE AML study. Patients considered Low Risk will receive the standard treatments outside of the UPDATE AML trial but will be eligible for the non-treatment parts of the trial. IR and HR patients will receive a combination of idarubicin, fludarabine, cytarabine (Ida-FLA) as their 2nd cycle of chemotherapy ("Induction 2"). This combination has shown desirable anti-leukemic activity in children whose leukemia has relapsed but has not yet been studied extensively in children newly diagnosed with AML. Secondly the trial will administer the new drug venetoclax (FDA approved for adults with AML but not for pediatric patients) combined with idarubicin and cytarabine as the 3rd or 4th cycle (of the HR or IR regimens respectively). Texas Children's Hospital will be providing the venetoclax.

The other major goal of UPDATE AML is to improve to detection of residual leukemia. Currently, the intensity of treatment for pediatric patients with AML depends on the genetic changes in the leukemia cells and their response to the first month of therapy. Of patients who have no detectable residual disease at the end of the first month, 30% of them will still relapse, indicating residual leukemia was still present, just not detected. Our study will develop individualized tests for each patient's genetic change which should increase detection of tiny amounts of residual leukemia. If our trial can successfully develop these individualized tests, future pediatric AML trials will incorporate these tests into use for all patients.

The research study procedures include screening for eligibility study treatment, evaluation, administration of the substituted chemotherapy cycles, and follow-up visits. Participants will be offered the possibility to provide additional blood and bone marrow samples (to be collected only at times of regular medical examination). There are additional surveys patients and parents can participate in, to understand the challenges facing families undergoing pediatric AML treatment.

Besides the 2 substituted chemotherapy cycles, patients will otherwise receive standard chemotherapy as their relapse risk indicates. Patients will be followed for approximately 3 years from enrollment.

It is expected that about 36 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

- Age Patients ≥ 1 months old to ≤ 30 years old are eligible

Patients must be diagnosed with AML or myeloid sarcoma according to the 2022 WHO classification with or without extramedullary disease. Patients with AML must have 1 of the following at initial diagnosis:

1. ≥ 20% bone marrow blasts

   • In cases where extensive fibrosis may result in a dry tap, blast count can be obtained from touch imprints or estimated from an adequate bone marrow core biopsy.
2. < 20% bone marrow blasts with one or more of the genetic abnormalities below:

   * t(8;21)(q22;q22.1) RUNX1::RUNX1T1
   * inv(16)(p13.1q22) or t(16;16)(p13.1;q22) CBFB::MYH11
   * Translocation involving 11q23.3 KMT2A rearrangement
   * t(6;9)(p23;q34.1) DEK::NUP214
   * inv(3)(q21.3q26.2) or t(3;3)(q21.3;q26.2) MECOM rearrangement
   * Megakaryoblastic with t(1;22)(p13.3;q13.3) RBM15::MRTFA
   * Mutated NPM1
   * t(5;11)(q35.3;p15.5) NUP98::NSD1
   * inv(16)(p13.3q24.3) CBFA2T3::GLIS2
   * t(11;12)(p15.5;p13.5) NUP98::KDM5A
3. A complete blood count (CBC) documenting the presence of at least 1,000/µL circulating leukemic cells (blasts) if a bone marrow aspirate or biopsy cannot be performed (i.e., a WBC count ≥ 10,000/μL with ≥ 10% blasts or a WBC count of ≥ 5,000/μL with ≥ 20% blasts).
4. Biopsy-proven myeloid sarcoma with or without bone marrow involvement.

   Note: patients with newly diagnosed AML, myelodysplasia-related (that are not from conditions listed in protocol section 4.2.1) ARE eligible while patients with therapy-related AML are excluded.

   Prior Therapy Patients must receive DA10+GO (Cytarabine days 1-10 + Daunorubicin days 1,3,5 [DA10] + Gemtuzumab ozogamcin [GO]) as prescribed in AAML1831 or the TXCH practice standard for Induction 1. Patients may have received any number of intrathecal treatments and have any CNS status at the time of enrollment.

   Performance Status Patients must have a performance status corresponding to Karnofsky/Lansky score >40. (Use Karnofsky for patients ≥16 years of age and Lanksy for patients <16 years of age.)

   Organ Function Requirements All laboratory studies to determine eligibility must be performed within 7 days prior to enrollment unless otherwise indicated. Laboratory values used to assess eligibility must be no older than seven (7) days at the start of therapy. Laboratory tests need not be repeated if therapy starts within seven (7) days of obtaining labs to assess eligibility. If a post-enrollment lab value is outside the limits of eligibility, or laboratory values are > seven (7) days old, then the following laboratory evaluations must be re-checked within 48 hours prior to initiating therapy: CBC with differential, bilirubin, ALT (SGPT) and serum creatinine. If the recheck is outside the limits of eligibility, the patient may not receive protocol therapy and will be considered off protocol therapy.

   Adequate renal function defined as:

   • A creatinine clearance or GFR ≥ 60 ml/min/1.73m2

   Adequate liver function defined as:

   • A direct bilirubin < 2 mg/dL

   • ALT <5x ULN or 225 U/L, with the ULN being 45 U/L for the purpose of this study.

   Adequate coagulation defined as:

   • INR ≤ 1.5

   Adequate cardiac function defined as:
   * Ejection fraction (EF) ≥ 50% (preferred method Biplane Simpson's EF) or if EF unavailable, shortening fraction (SF) ≥ 24%, within 14 days prior to planned start of Induction 2 therapy.
   * For patients with cardiac dysfunction (EF < 50% or SF <24% if EF is unavailable) prior to enrollment, if clinically safe and feasible, repeat echocardiogram is strongly advised in order to confirm cardiac dysfunction following clinical stabilization, particularly if occurring in the setting of sepsis or other transient physiologic stressor. If the repeat echocardiogram demonstrates an EF ≥ 50%, the patient is eligible to enroll.

   Informed Consent All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.

   Exclusion Criteria:

   - Patients with the following constitutional conditions are not eligible:

   • Fanconi anemia

   • Schwachman Diamond Syndrome

   • Telomere Disorders

   • Patients with constitutional trisomy 21 or with constitutional mosaicism of trisomy 21

   • Germline predispositions known, or suspected by the treating physician, to increase risk of toxicity with AML therapy
   * Therapy-related AML

   Patients with any of the following oncologic diagnoses are not eligible:

   • Any concurrent malignancy

   • Juvenile myelomonocytic leukemia

   • Philadelphia chromosome positive AML
   * Mixed phenotype acute leukemia
   * Acute promyelocytic leukemia
   * AML with FLT3 internal tandem duplication (FLT3-ITD)

   Pregnancy and Breastfeeding
   * Female patients who are pregnant may not participate. A pregnancy test is required for female patients of childbearing potential.
   * Lactating females who plan to breastfeed their infants are not eligible.
   * Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation are not eligible.

Ages: 1 Month to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
Tolerability rate of Ida-FLA | From Day 1 of Ida-FLA through up to 50 days after completion of Ida-FLA
  Tolerability rate is the proportion of participants in the tolerability dataset who did not experience an intolerable event during Induction 2 for IR and HR patients. Number of intolerable participants will be used. Intolerability is defined by events outlined in Section 6.6 of the protocol as follow:
  Non-Hematological Toxicity: Any Grade 5 toxicity, Grade 4 cardiac disorder, Grade 4 infection, or other Grade 4+ non-hematologic toxicity except:
  * Grade 4 nausea/vomiting (<3 days)
  * Grade 4 ALT/AST/GGT elevation (returns to ≤Grade 1 before next cycle)
  * Grade 4 electrolyte abnormalities (corrected by supplementation)
  * Cycle delays >50 days indicate intolerability. Hematologic Toxicity: Intolerability includes failure to recover ANC >500/mL and platelets >20,000/mL (without transfusion in past 7 days) by day 50 or cycle start delay >50 days.
  A cycle of Ida-FLA is 29-56 days.
Tolerability rate of VIA for IR patients | From Day 1 of VIA through up to 50 days after completion of VIA
  Tolerability rate is the proportion of participants in the tolerability dataset who did not experience an intolerable event during intensification 2 for IR patients as the 4th cycle. Number of intolerable participants will be used. Intolerability is defined by events outlined in Section 6.6 of the protocol as follow:
  Non-Hematological Toxicity: Any Grade 5 toxicity, Grade 4 cardiac disorder, Grade 4 infection, or other Grade 4+ non-hematologic toxicity except:
  * Grade 4 nausea/vomiting (<3 days)
  * Grade 4 ALT/AST/GGT elevation (returns to ≤Grade 1 before next cycle)
  * Grade 4 electrolyte abnormalities (corrected by supplementation)
  * Cycle delays >50 days indicate intolerability. Hematologic Toxicity: Intolerability includes failure to recover ANC >500/mL and platelets >20,000/mL (without transfusion in past 7 days) by day 50 or cycle start delay >50 days.
  A cycle of VIA is 29-56 days.
Tolerability rate of VIA for HR patients | From Day 1 of VIA through up to 50 days after completion of VIA
  Tolerability rate is the proportion of participants in the tolerability dataset who did not experience an intolerable event during intensification 2 for HR patients as the 3rd cycle. Number of intolerable participants will be used. Intolerability is defined by events outlined in Section 6.6 of the protocol as follow:
  Non-Hematological Toxicity: Any Grade 5 toxicity, Grade 4 cardiac disorder, Grade 4 infection, or other Grade 4+ non-hematologic toxicity except:
  * Grade 4 nausea/vomiting (<3 days)
  * Grade 4 ALT/AST/GGT elevation (returns to ≤Grade 1 before next cycle)
  * Grade 4 electrolyte abnormalities (corrected by supplementation)
  * Cycle delays >50 days indicate intolerability. Hematologic Toxicity: Intolerability includes failure to recover ANC >500/mL and platelets >20,000/mL (without transfusion in past 7 days) by day 50 or cycle start delay >50 days.
  A cycle of VIA is 29-56 days.

SECONDARY OUTCOMES:
Complete remission rate | at the end of Induction 2 which may occur between day 29 and day 56 of the cycle
  Complete remission (CR/CRi/CRp) will be defined asbone marrow blast <5% by morphology with regenerating normal hematopoietic cells, negative CSF cytology, and no extramedullary disease. Number of complete remission respondents.The complete remission rate will be estimated as the proportion of the Induction 2 population that is in complete remission at the end of Induction 2 for IR and HR patients A cycle of Ida-FLA(induction 2) is 29-56 days.
MRD negative rate | at the end of Induction 2 which may occur between day 29 and day 56 of the cycle
  The MRD assessment will be based on the subset of the Induction 2 in IR + HR population that were MRD positive at the end of Induction 1.The MRD negative rate will be estimated as the proportion of IR+HR patients who are MRD negative (<0.05% by flow cytometry) at the end of Induction 2, out of the number of IR+HR patients who were MRD positive (>0.05% by flow cytometry) at the end of Induction 1.
  A cycle of Ida-FLA(induction 2) is 29-56 days.
3 year event-free survival | from enrollment up to 3 years
  Event-free survival (EFS) is defined as the time from study enrollment until refractory disease or relapse, death due to any cause or last date of follow-up over 3 years in IR and HR, separately. The median survival time will be estimated using the Kaplan-Meier method.
3 year overall survival | From enrollment up to 3 years
  Overall survival (OS) is defined as time from study entry until death due to any cause or last date of follow-up over 3 years in IR and HR, separately.The median survival time will be estimated using the Kaplan-Meier method.
Rate of count recovery in IR Intensification 1 | at the end of Intensification 1 which may occur between day 29 and day 56 of the cycle
  The time to post-nadir recovery of absolute neutrophil count (ANC) to >500/μL and platelets to >20,000/μL (without transfusion) is determined for IR patients at the end of Intensification 1. Count recovery is defined above. Day 42 is a standard benchmark for count recovery, beyond which recovery is considered delayed. The proportion of IR patients who achieve full count recovery by day 42 of Intensification 1 will be estimated using the Kaplan-Meier method.
  A cycle of intensification 1 is 29-56 days.
Tolerability rate of intensified regimen as a whole for IR patients | at the end of Intensification 3 which may occur between day 29 and day 56 of the cycle
  Tolerability of the IR regimen overall is assessed at the end of Intensification 3 for IR patients.
  The overall tolerability rate for IR patients receiving the intensified IR regimen as a whole will be calculated as the proportion of IR patients who complete of protocol therapy without severe toxicity requiring removal from the regimen, as defined in Section 6.6 of the protocol as follow:
  Non-Hematological Toxicity: Any Grade 5 toxicity, Grade 4 cardiac disorder, Grade 4 infection, or other Grade 4+ non-hematologic toxicity except:
  * Grade 4 nausea/vomiting (<3 days)
  * Grade 4 ALT/AST/GGT elevation (returns to ≤Grade 1 before next cycle)
  * Grade 4 electrolyte abnormalities (corrected by supplementation)
  * Cycle delays >50 days indicate intolerability. Hematologic Toxicity: Intolerability includes failure to recover ANC >500/mL and platelets >20,000/mL (without transfusion in past 7 days) by day 50 or cycle start delay >50 days.
  A cycle of intensification 3 is 29-56 days.
Tolerability rate of intensified regimen as a whole for HR patients | at day 30 after completion of HSCT
  Tolerability of the HR regimen overall is assessed at day +30 after HSCT for HR patients.
  The overall tolerability rate for HR patients receiving the intensified HR regimen as a whole will be calculated as the proportion of HR patients who complete of protocol therapy and HSCT without severe toxicity requiring removal from the regimen, as defined in Section 6.6 of the protocol as follow:
  Non-Hematological Toxicity: Any Grade 5 toxicity, Grade 4 cardiac disorder, Grade 4 infection, or other Grade 4+ non-hematologic toxicity except:
  * Grade 4 nausea/vomiting (<3 days)
  * Grade 4 ALT/AST/GGT elevation (returns to ≤Grade 1 before next cycle)
  * Grade 4 electrolyte abnormalities (corrected by supplementation)
  * Cycle delays >50 days indicate intolerability. Hematologic Toxicity: Intolerability includes failure to recover ANC >500/mL and platelets >20,000/mL (without transfusion in past 7 days) by day 50 or cycle start delay >50 days..
  A cycle is 29-56 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Children's Cancer and Hematology Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
All of the planned analyses, including the correlative biology, will be done by members of the study committee.